CLINICAL TRIAL: NCT02516618
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of Fasinumab in Healthy Japanese and Caucasian Subjects
Brief Title: Study of Fasinumab (REGN475) in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R475-PN-1516
Record Dates: First submitted 2015-07-31; First posted 2015-08-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): Participants in this cohort will receive dose 1 of Fasinumab or placebo
  Interventions: Drug: Fasinumab; Drug: Placebo
- Cohort 2 (Experimental): Participants in this cohort will receive dose 2 of Fasinumab or placebo
  Interventions: Drug: Fasinumab; Drug: Placebo
- Cohort 3 (Experimental): Participants in this cohort will receive dose 3 of Fasinumab or placebo
  Interventions: Drug: Fasinumab; Drug: Placebo
- Cohort 4 (Experimental): Participants in this cohort will receive dose 4 of Fasinumab or placebo
  Interventions: Drug: Fasinumab; Drug: Placebo
- Cohort 5 (Experimental): Participants in this cohort will receive dose 5 of Fasinumab or placebo
  Interventions: Drug: Fasinumab; Drug: Placebo

INTERVENTIONS:
Drug: Fasinumab
  Other Names: REGN475
Drug: Placebo

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of a single dose of subcutaneous (SC) or intravenous (IV) administered fasinumab in healthy Japanese subjects.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male or female Japanese and Caucasian volunteers ≥20 and ≤55 years of age at the screening visit
2. Japanese subjects must:

   * Be first generation Japanese, defined as born in Japan and having 4 biologic grandparents who are ethnic Japanese
   * Have maintained a Japanese lifestyle since leaving Japan
3. Caucasian subjects must be Caucasian of European or Latin American descent
4. Have a Body Mass Index (BMI) ≤ 35
5. Be willing to refrain from taking NSAID medications (oral or topical) for 1 week prior to receiving study drug and for 16 weeks after study drug administration

Key Exclusion Criteria:

1. History or presence at the screening visit of bone or joint disorders including but not limited to osteoarthritis, avascular necrosis, destructive arthropathy, pathologic fractures, osteonecrosis, rheumatoid arthritis, neuropathic joint arthropathy, lupus erythematosus, or inflammatory joint diseases
2. History of joint-related events such as, but not limited to, total joint replacement (TJR) surgery, patella dislocation, hip dislocation, knee dislocation, injury to meniscus or knee ligaments (with or without surgical repair), or joint infections
3. Trauma to any joint in the 30 days prior to the screening visit
4. History of autonomic neuropathy, or diabetic neuropathy
5. Evidence of autonomic neuropathy
6. Presence of clinically relevant peripheral neuropathy
7. History or presence at the screening visit of orthostatic hypotension
8. History or evidence at screening of heart block
9. Resting heart rate of <50 or >100 beats per minute (bpm)
10. History of poorly controlled hypertension:
11. Congestive heart failure with NY Heart Classification of stage 3 or 4
12. History of myocardial infarction, acute coronary syndromes, or cerebrovascular accident within 12 months prior to the screening visit
13. Significant concomitant illness such as, but not limited to, cardiac, renal, neurological, endocrinological, GI, hepatic, metabolic or lymphatic disease that would adversely affect the subject's participation in this study or interpretation of safety/PK data
14. HIV, hepatitis B, or hepatitis C positive by serological testing at the screening visit
15. History or presence of malignancy within 5 years prior to screening, except subjects who have been treated successfully with no recurrence of basal or squamous cell carcinoma of the skin (< 1 year), in situ cervical cancer, or in situ ductal breast cancer
16. Women of reproductive potential who have a positive serum pregnancy test result at the screening visit, or a positive urine pregnancy test result at the baseline visit, or who do not have their pregnancy test results at the baseline visit
17. Pregnant or breast-feeding women
18. Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives of the investigational drug, whichever is longer, prior to the day 1 visit

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in the study is the incidence and severity of treatment emergent adverse events (TEAEs) in participants treated with fasinumab or placebo. | Baseline to week 16 (End of Study)

SECONDARY OUTCOMES:
Fasinumab serum concentrations over time | Baseline to week 16 (End of Study)
Presence of anti-fasinumab antibodies over time | Baseline to week 16 (End of Study)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Glendale, California, United States